CLINICAL TRIAL: NCT03724019
Title: Evaluation of the Impact of the Use of Ketamine in Laparoscopic Surgery, Using the Quality of Recovery 15 Questionnaire.
Brief Title: Impact of the Use of Ketamine in Laparoscopic Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: QuetaminaQOR15
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-09

CONDITIONS: Quality of Recovery
Keywords: Ketamine; QoR-15; Laparoscopic surgery
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group Q (Experimental): 20 milliliter of ketamine (0.5mg / kg ideal body weight) at induction of anesthesia.
  Interventions: Drug: Ketamine
- Group S (No Intervention)

INTERVENTIONS:
Drug: Ketamine — Administration of 0.5mg / kg ideal body weight of ketamine at induction of anesthesia in laparoscopic surgery.
  Arms: Group Q

SUMMARY:
In order to improve the postoperative period (namely pain control), several drugs can be used. For instance, ketamine is a general anesthetic that holds strong analgesic properties, yet also owns undesirable effects, in which hallucination phenomena is one the most common indicator. However, slight information is available about the real implication in the quality of the recovery on the use of ketamine for postoperative pain treatment. The quality of the recovery includes several health conditions, such as pain, physical comfort, physical independence, psychological support and emotional state. In recent years, investigations in this field has been attracted the attention by the health professionals, since is an indicator of the quality of post-operative care. To evaluate these parameters, questionnaires have been developed, in which the Portuguese version of Quality of Recovery 15 (QoR-15) is include. This questionnaire evaluates five psychometric dimensions. Therefore, the present study has the main goal, the evaluation of the effect of using ketamine in laparoscopic surgery and the quality of the recovery using the QoR-15 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years age, with an American Society of Anesthesiology physical status I, II or III.
* Laparoscopic surgery (sleeve gastrectomy, salpingectomy, or cholecystectomy)

Exclusion Criteria:

* patient refusal, the incapacity of providing informed consent, drug abusers (current or past history) or alcohol abuse, medication with benzodiazepines, inability to give informed consent, pregnant, emergency surgery, psychiatric pathology, existence of surgical complications in the recovery and admission to a level II or III unit ( for any reason).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Impact in QoR-15 score | 6 months
  Difference (improvement or worsening) in the postoperative baseline score (preoperative) in the Portuguese version of the Quality of Recovery questionnaire 15.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU São João, Porto, Portugal

REFERENCES:
- [Derived] Pereira H, Graca MI, Fonseca D, Mendes-Castro A, Abelha F. Impact of Ketamine on Quality of Recovery after Laparoscopic Surgery: A Single-Centre Single-Blinded Trial Using the QoR-15 Questionnaire. Anesthesiol Res Pract. 2023 Jan 20;2023:8890025. doi: 10.1155/2023/8890025. eCollection 2023. PMID 36714040